CLINICAL TRIAL: NCT04569682
Title: Outcomes of Transrenal Artery Perfusion Versus Transrenal Vein Perfusion Using LifePort for Deceased Donor Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Tao Lin, Deputy Director of the Organ Transplant Center, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: WestChina-LifePort
Record Dates: First submitted 2020-09-21; First posted 2020-09-30 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Kidney Transplantation; Organ Preservation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transrenal artery perfusion group (Active Comparator)
  Interventions: Device: LifePort transrenal artery perfusion
- transrenal vein perfusion group (Experimental)
  Interventions: Device: LifePort transrenal vein perfusion

INTERVENTIONS:
Device: LifePort transrenal artery perfusion — transrenal artery perfusion group
  Arms: transrenal artery perfusion group
Device: LifePort transrenal vein perfusion — transrenal vein perfusion group
  Arms: transrenal vein perfusion group

SUMMARY:
The main objective of this study is to compare the outcomes of transrenal artery perfusion versus transrenal vein perfusion using LifePort for deceased donor kidney transplantation. Patients registered in the National Dialysis and Transplant Registry awaiting deceased donor kidney transplantation were included. Delayed graft function (DGF) or primary nonfunction (PNF) may occur after deceased donor kidney transplantation. Compared with static cold storage, the application of LifePort can significantly reduce the incidence of DGF and PNF in deceased donor kidney transplantation. Transrenal artery perfusion is currently the mainstream but confronts multiple renal arteries, resulted in prolonged cold ischemia time. Transrenal vein perfusion is expected to be a solution. However, whether the clinical outcomes of transrenal vein perfusion is inferior to transrenal artery perfusion remains unknown. In this study, values of urine volume and creatinine, incidence and duration of DGF, and incidence of PNF within 1 week after surgery are recorded and compared between the transrenal artery perfusion group and the transrenal vein perfusion group. Monthly eGFR and creatinine values, the incidence of acute rejection within 1 year after transplantation and 1-year graft and patient survival are also recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Adult recipients older than 18 years;
2. Patients diagnosed with end-stage renal diseases and volunteered to register in the Transplant and Dialysis Registry of China awaiting for deceased donor kidney transplantation;
3. First single kidney transplantation;
4. The recipients can understand the purpose and risk of deceased kidney transplantation and sign informed consent;
5. Ethics committee approved.

Exclusion Criteria:

1. Patients less than 18 years old, or more than 65 years old;
2. Patients who receive multiple organ transplants;
3. Diagnosed with malignancy or had a history of malignancy in the past 5 years;
4. non-kidney transplantation history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Delayed graft function | Within one week posttransplantation
  Delayed graft function is defined as the need for dialysis (for any cause) within the first week posttransplantation.

SECONDARY OUTCOMES:
Graft loss | One year after transplantation
  Graft loss was defined as re-establishment of long-term dialysis or estimated glomerular filtration rate (eGFR) of <15 ml/min.
biopsy-confirmed acute rejection | One year after transplantation
  biopsy-confirmed acute rejection was diagnosed clinically based on a significant increase in serum creatinine levels of 50% or more within 3 days, which was not explained by other reasons and confirmed by biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743
- [Derived] Zhang H, Zeng J, Fan Y, Ma M, Lin T, Song T. Continuous renal surface cooling technique (CSCT) in robotic-assisted kidney transplantation: technique and outcomes from a high-volume center: a prospective cohort study. Int J Surg. 2024 Jul 1;110(7):4143-4150. doi: 10.1097/JS9.0000000000001385. PMID 38742842